CLINICAL TRIAL: NCT02195115
Title: Randomized Controlled Trial of Laparoscopic Cholecystectomy vs. Non-operative Treatment for Gallbladder Dyskinesia
Brief Title: Trial of Laparoscopic Cholecystectomy vs. Non-operative Treatment for Gallbladder Dyskinesia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CAMC Health System (Other)
Collaborators: University of Kentucky (Other); National Center for Research Resources (NCRR) (NIH); National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ULJRR033173; U54GM104942 (NIH)
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2014-07

CONDITIONS: Gallbladder Dyskinesia
MeSH Terms: conditions — Biliary Dyskinesia | interventions — Cholecystectomy, Laparoscopic; Amitriptyline; Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic cholecystectomy (Active Comparator): surgical removal of gallbladder
  Interventions: Procedure: Laparoscopic Cholecystectomy
- Non-operative treatment (Active Comparator): Administration of amitriptyline 25mg daily, Low Fat-Low Cholesterol Diet
  Interventions: Drug: amitriptyline; Other: low-fat and low cholesterol diet

INTERVENTIONS:
Procedure: Laparoscopic Cholecystectomy
  Arms: Laparoscopic cholecystectomy
Drug: amitriptyline
  Arms: Non-operative treatment
Other: low-fat and low cholesterol diet
  Arms: Non-operative treatment

SUMMARY:
The goal of this study is to challenge the existing clinical practice of employing laparoscopic cholecystectomy as the treatment for gallbladder dyskinesia by comparing it to a regimen of active non-surgical therapy.

DETAILED DESCRIPTION:
Willing and eligible patients will be enrolled into the trial and randomized to surgical vs non-surgical treatment following informed consent. The following information will be collected over the next 18 months: age,race, sex, baseline and follow-up quality of life quationnaire scores, a complete medical history, including co-morbid illnesses, medications and surgical history, and a complete assessment of symptoms, including disease specific symptoms against the Rome III criteria for functional gallbladder disorder. Patients randomized to surgery will be referred for immediate laparoscopic cholecystectomy. Patients in the non-surgical management group will be counseled on maintenance of a low-fat diet, and provided with a prescription for amitriptyline 25mg once daily.

Patients with persistent, non responsive symptoms that fail to respond to at least one week of administration of amitriptyline will be allowed to voluntarily, cross over into the surgically treated group.

After randomization, certain data collection points will be unique to the two groups. These are as follows and are in addition to the general data which will be collected from both groups:

Surgery group: operative/pathology findings & operative complications

Non-surgical group:

Patients will be asked to maintain a food diary and a symptom diary. Patients will be asked to report any medication related side effects.

Both groups will receive a phone call for assessment of conditions. Non-surgical groups will be asked to report any medication related side effects.

Follow-up for both groups will continue throughout the 18 month period. In addition to the monthly calls, Patients will be contacted every three months after their initial treatment to take the SF-8 questionnaire and obtain an assessment of symptoms using the Rome III criteria.

ELIGIBILITY:
Inclusion Criteria:

Patients with a normal gallbladder Patients with symptoms compatible with gallbladder dyskinesia (functional gallbladder disorder) as defined by the Rome III criteria Patients with a Cholecystokinin hepatobiliary (CCK-HIDA) scintigraphy gallbladder ejection fraction of <38%, performed at a facility using updated Society of Nuclear Medicaine guidelines for test administration

Exclusion Criteria:

Patients with other known sources of chronic abdominal pain (ex: Crohn's disease) Patients with chronic narcotic use which will affect the reproducibility and validity of the CCK-HIDA results Patient with a history of allergy to amitriptyline Patients with a seizure disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
SF-8 | 18 months
  Administration of SF-8 (health questionnaire) survey prior to the initiation of treatment and periodically after the initiation of treatment to assess the ability of cholecystectomy to provide durable symptomatic relief.

SECONDARY OUTCOMES:
Rome III Criteria | 18 months
  Comparison of the results of surgery to those of non-surgical treatment based on degree of relief of symptoms described in the Rome III criteria and follow-up SF-8 scores.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan K Richmond, MD, Principal Investigator — West Virginia University, Charleston Division ; Professor of Surgery
Locations (1):
- Charleston Area Medical Center, Charleston, West Virginia, United States